CLINICAL TRIAL: NCT01200823
Title: Collection of Blood, Bone Marrow, Leukapheresis, and Tissue Biopsy Samples From Patients and Their Family Members for Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI) Laboratory Research Studies
Brief Title: Collection of Blood, Bone Marrow, Leukapheresis, and Tissue Biopsy Samples From Patients and Their Family Members for Center for Human Immunology, Autoimmunity, and Inflammatory Diseases Laboratory Research Studies
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100162; 10-I-0162
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09-18

CONDITIONS: Idopathic Inflammatory/Autoimmune Syndromes
Keywords: Laboratory Research; Biologic Samples; Tissue Collection; Tissue Procurement

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

- The Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI) is conducting a variety of laboratory research experiments that require blood, bone marrow, urine, stool, and/or tissue samples from patients with a diagnosis of an immunologic, autoimmune, or inflammatory disorder, as well as from their healthy relatives. Donated samples will be sent to the CHI laboratory at the National Institutes of Health to be used in research that may provide more information on the changes in the immune system caused by these specific disorders.

Objectives:

- To collect blood, leukapheresis cells, bone marrow, urine, stool, cheek swab, and tissue samples from patients with immune-mediated and inflammatory diseases, as well as from family members, for ongoing exploratory research studies.

Eligibility:

* Individuals at least 2 years of age who have been diagnosed with an immune-mediated or inflammatory disease, or have signs or symptoms of an immune or inflammatory disease without a formal diagnosis.
* Immediate family members (parent, child, sibling, grandchild) of the above mentioned individuals.

Design:

* Participants will be screened with a complete medical history, physical examination, and blood and urine samples.
* Participants will provide blood, urine, stool, cheek swab, and tissue samples as required by the study researchers.
* Participants who have immune or inflammatory diseases will also provide blood and bone marrow samples collected through biopsies and leukapheresis (to collect specific blood cells).
* Adult relatives will provide additional samples through more invasive procedures such as leukapheresis and bone marrow biopsies. Child relatives (between 2 and 18 years of age) will not undergo these invasive procedures.
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
BACKGROUND

Clinical investigators in the Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI) study the pathophysiology of a wide variety of immune-mediated and inflammatory diseases. One of the goals of the CHI is to better understand these diseases and to refine therapeutic approaches used in their management based on knowledge of the underlying pathophysiologies. This requires samples from patients with immune-mediated and inflammatory diseases for such clinical and laboratory assessments. Collection of samples from family members is necessary to identify genetic components of specific conditions.

We expect the great majority of publications from the Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI) over the next several decades will be generated from exploratory laboratory research studies done using blood and bone marrow and other tissue samples from such patients and their family members. These publications are expected to number in the hundreds. Ongoing and future research projects depend on the ready availability of samples of blood, tissue, leukapheresed cells, and bone marrow from patients for in vitro studies.

OBJECTIVE

To provide a mechanism for collection of blood, bone marrow, leukapheresis cells, urine, stool, buccal mucosa and/or tissue samples from patients with immune-mediated and inflammatory diseases, as well as from family members for ongoing exploratory research studies.

STUDY DESIGN

This study is not a treatment protocol. This is a sample and clinical data procurement protocol.

All subjects with conditions of interest seen at the NIH Clinical Center will first be enrolled onto CHI protocol 09-H-0201 Screening protocol for subjects being evaluated for Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI) protocols. Patients who require specific medical intervention will be enrolled on and receive treatment under another NIH or CHI Clinical Center protocol or will be under the care of their home health care provider. In exceptional cases in which it is not possible for patients to travel to the Clinical Center, they may be allowed the option of giving consent to provide samples for research studies, including genetic analyses, performed on blood, buccal mucosa, bone marrow, and tissue samples sent through their local physician without enrolling onto 09-H-0201. Information will be obtained retrospectively by review of medical records and examination of archived materials and/or prospectively by clinical examinations and laboratory tests. The protocol is written for an indefinite period of time with subject accrual to occur both at the NIH Clinical Center or through home health care providers (off site).

ELIGIBILITY:
* INCLUSION CRITERIA

Affected Adults

* The subject carries the diagnosis of an immune-mediated or inflammatory disease, or has signs or symptoms of an immune or inflammatory disease without a formal diagnosis.
* Age 18 years and older (no upper limit)

Affected Children

* The subject carries the diagnosis of an immune-mediated or inflammatory disease, or has signs or symptoms of an immune or inflammatory disease without a formal diagnosis.
* Age 2 years and older (no upper limit)

Unaffected Child Relatives

* Immediate family members (child, sibling, grandchild) of individuals included under item (Affected Adult)
* Subjects over 2 years of age may (but < 18 years of age) be seen for initial evaluations, genetic studies, or research blood specimens, or may send blood or buccal samples for genetic testing only. Unaffected family members will not be asked to undergo leukapheresis, bone marrow aspirations and biopsies, or other invasive procedures.

Unaffected Adult Relatives

* Immediate family members (parent, child, sibling, grandchild) of individuals included under item (Affected Adult)
* Subjects over 18 years of age may be seen for initial evaluations, genetic studies, or research blood specimens, or may send blood or buccal samples for genetic testing only. Unaffected family members will not be asked to undergo leukapheresis, bone marrow aspirations and biopsies, or other invasive procedures.

EXCLUSION CRITERIA: (All groups)

* Subjects or their parents or guardians who are unable to comprehend the investigational nature of the procedure. The subject or the subject s guardian is unable to understand the investigational nature of the study and provide informed consent after initial counseling by clinical staff. Only adults capable of signing consent will be eligible. Separate consent forms for all interventional or surgical procedures will be obtained after explanation of the specific procedure.
* Pregnant unaffected relatives will be excluded.
* Subjects not willing to participate in the genetic analysis and whole genomic analysis portion of this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-07-01; Study Completion 2018-09-18

PRIMARY OUTCOMES:
Samples will be used for clinical and translational research in the CHI and are indispensable for many of our research projects, including understanding the pathophysiology of a wide variety of immune-mediated and inflammatory diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Biancotto, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cole M, Boddy AV, Kearns P, Teh KH, Price L, Parry A, Pearson AD, Veal GJ; UKCCSG Pharmacology group. Potential clinical impact of taking multiple blood samples for research studies in paediatric oncology: how much do we really know? Pediatr Blood Cancer. 2006 Jun;46(7):723-7. doi: 10.1002/pbc.20463. PMID 16007598
- [Background] Wood AJ, Darbyshire J. Injury to research volunteers--the clinical-research nightmare. N Engl J Med. 2006 May 4;354(18):1869-71. doi: 10.1056/NEJMp068082. No abstract available. PMID 16672696
- [Background] Wolthers OD. A questionnaire on factors influencing children's assent and dissent to non-therapeutic research. J Med Ethics. 2006 May;32(5):292-7. doi: 10.1136/jme.2004.010579. PMID 16648281
- [Derived] El-Chemaly S, Cheung F, Kotliarov Y, O'Brien KJ, Gahl WA, Chen J, Perl SY, Biancotto A, Gochuico BR. The Immunome in Two Inherited Forms of Pulmonary Fibrosis. Front Immunol. 2018 Jan 31;9:76. doi: 10.3389/fimmu.2018.00076. eCollection 2018. PMID 29445374